CLINICAL TRIAL: NCT06723548
Title: The Efficacy and Safety of Telitacicept Combined With Low-dose Steroids in Patients With Refractory Myasthenia Gravis
Brief Title: Telitacicept and Low-dose Steroids in Refractory Myasthenia Gravis
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: First Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-ps-195
Record Dates: First submitted 2024-11-15; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-11

CONDITIONS: Myasthenia Gravis; Autoimmune Diseases
MeSH Terms: conditions — Myasthenia Gravis; Autoimmune Diseases | interventions — telitacicept; Pyridostigmine Bromide; Prednisone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with refractory MG treated with Telitacicept combined with low-dose steroids (Experimental): This is an open-label, single-arm exploratory study of Telitacicept (240mg weekly, then every two weeks after achieving MMS or QMG reduction of ≥ 6 points) combined with a gradual reduction of steroids and other immunosuppressants. When the steroid dose is reduced to 5mg/day or 10mg/every other day, Telitacicept can be reduced to 160mg, administered subcutaneously every two weeks.
  Interventions: Drug: Telitacicept

INTERVENTIONS:
Drug: Telitacicept — Patients with MG who fulfill the inclusion criteria will receive Telitacicept 240mg weekly as an adjunct to their medication. Upon reaching MMS, significant symptom improvement, or a QMG score reduction of at least 6 points, Telitacicept is reduced to biweekly doses. Pyridostigmine and NSISTs are tapered based on patient response. Following this, Prednisone is tapered, starting with rapid reduction early and slowing later. If a patient on 60mg Prednisone daily achieves treatment goals within 6-8 weeks of Telitacicept initiation, the tapering sequence is 60mg every other day for 4 weeks, then 30mg daily for 2-4 weeks, and so on, until reaching 5mg daily or 10mg every other day. At this point, Telitacicept may be reduced to 160mg biweekly.
  Other Names: Pyridostigmine Bromide; NSISTs; prednisone

SUMMARY:
This study is designed to explore the efficacy and safety of Telitacicept combined with low-dose steroids for the treatment of refractory MG, and to investigate related biomarkers such as immunoglobulins, BlyS/APRIL, and AChR-Ab titers, in order to clarify whether Telitacicept can rapidly and effectively help achieve MG treatment goals and assist in steroid reduction.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-85 years, both genders included；
* Meet the diagnostic criteria of the 2020 Chinese MG guidelines, with positive serological testing for AChR-Ab;
* Clinical classification of Type I to Type IVa according to the MGFA;
* Meet the criteria for refractory MG in the 2022 Japanese MG guidelines: poor response to standard treatment, intolerance to standard treatment drugs due to adverse reactions, frequent relapses/exacerbations after reduction of standard treatment drugs, frequent need for rescue treatment due to disease fluctuations, frequent myasthenic crises, and comorbidities that limit the use of standard treatment;
* Patients with unstable symptoms (MG-ADL score ≥6 or QMG ≥8) despite treatment with standard therapeutic regimens before enrollment, defined as follows:

  1. Patients on monotherapy with corticosteroids: a corticosteroid dose ≤60mg/d, and a stable dose for at least 1 month before enrollment;
  2. Patients on combination therapy with corticosteroids and other immunosuppressants: a corticosteroid dose ≤60mg/d, and a stable dose for at least 1 month before enrollment, while other immunosuppressants such as azathioprine, methotrexate, tacrolimus, and mycophenolate mofetil have been stable for 6 months prior to the study start and will remain stable during the study period;
* Patients must provide written informed consent.

Exclusion Criteria:

* Patients with active infections, such as herpes zoster, HIV, active pulmonary tuberculosis, or active hepatitis;
* Patients with thymic tumors or those who have undergone thymectomy within the past 6 months;
* Patients with coexisting malignant tumors;
* Patients with severe hepatic or renal insufficiency;
* Patients who have received intravenous immunoglobulin or undergone plasmapheresis within the last 2 months;
* Patients who have received any live vaccines within the last 3 months or plan to receive any vaccines during the study period;
* Women who are currently pregnant or breastfeeding, and patients who plan to conceive during the trial period;
* Patients with allergies to human-derived biological products;
* Patients who have participated in any clinical trial within the last 28 days or within 5 half-lives of the study medication (whichever is longer);
* Any other patients deemed unsuitable for enrollment by the investigator (e.g., severe psychiatric disorders).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The change in patients' ADL scores | from baseline to week 52
  The variation in ADL scores at 52 weeks compared to baseline in patients. Total MG -ADL scores range from 0 (normal) to 24 (severe).
The change in patients' QMG scores | from baseline to week 52
  The variation in QMG scores at 52 weeks compared to baseline in patients. Total QMG scores range from 0 (none) to 39 (severe).

SECONDARY OUTCOMES:
MGFA-PIS | from baseline to week 52
  Change in MGFA-PIS grading from baseline to week 52
the average daily corticosteroid usage | from baseline to week 24；from baseline to week 52
  Change in the average daily corticosteroid usage from baseline to week 24 during follow-up；Change in the average daily corticosteroid usage from baseline to week 52 during follow-up
the usage of traditional non-steroidal immunosuppressants | from baseline at weeks 24 and 52
  Change in the usage of traditional non-steroidal immunosuppressants from baseline to week 24 during follow-up; Change in the usage of traditional non-steroidal immunosuppressants from baseline to week 52 during follow-up. Medication usage logs or medical record reviews to document the changes in the use of traditional non-steroidal immunosuppressants (such as Azathioprine, Mycophenolate Mofetil, Tacrolimus, Methotrexate, Cyclosporine, etc.) from baseline to week 52. The change in the use of traditional non-steroidal immunosuppressants will be assessed by comparing the medication usage at baseline and at weeks 24 and 52. This includes details on the type of medication, dosage, frequency, and any adjustments or discontinuations.
Number of relapses | week 52
  Number of relapses in both groups by the end of treatment (clinical relapse is defined as an increase in QMG score of ≥3 points);
AUDTC | week 52
  Area under the corticosteroid dose-time curve (AUDTC) at week 52
Proportion of patients with a corticosteroid dose ≤10mg/d | at weeks 24 and 52
  Proportion of patients with a corticosteroid dose ≤10mg/d at weeks 24 and 52 during follow-up;
Proportion of patients achieving MMS with a corticosteroid dose ≤ 5mg/d | week 24
  Proportion of patients achieving MMS with a corticosteroid dose ≤5mg/d at week 24;
MG QoL15r scores | from baseline at weeks 24 and 52
  Change in MG QoL15r scores from baseline at weeks 24 and 52 during follow-up
safety（Incidence, severity, and outcome of adverse events） | 52 weeks
  Incidence, severity, and outcome of adverse events
relevant biomarkers | from baseline at week 52
  relevant biomarkers, such as immunoglobulins,lymphocyte subpopulation changes, BlyS/APRIL, and AChR-Ab titers.

IPD SHARING:
Plan to Share IPD: No